CLINICAL TRIAL: NCT06175533
Title: Decrease in Pain Score After Ultrasound Guided CRF for Chronic Plantar Fasciitis Not Responding to Treatment in Addition to Ultrasound Changes
Brief Title: Pain Improvement After Ultrasound Guided Continuous Radio Frequency 60 Degree for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iraqi Board of medical specialties (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAQI BOARD
Record Dates: First submitted 2023-11-22; First posted 2023-12-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Intervention Model Description: chronic plantar fasciitis not responding to classical injection by steroid or regenerative therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plantar fasciitis (Experimental)
  Interventions: Procedure: ultrasound guided 60 degree CRF for plantar fasciitis

INTERVENTIONS:
Procedure: ultrasound guided 60 degree CRF for plantar fasciitis — ultrasound guided plantar fascia CRF for chronic conditions not responding to treatment

SUMMARY:
detailed changes after ultrasound guided cry for plantar fasciitis in regard pain score and plantar fascia AP diameter in ultrasound scan pre and 30 days post operation

ELIGIBILITY:
Inclusion Criteria:

* chronic plantar fasciitis not responding to treatment not responding to classical injection

Exclusion Criteria:

* torn plantar fascia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
reduction in pain score | 6 months
  reduction in pain score immediate and 1 week and 2 month according to NAS

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided